CLINICAL TRIAL: NCT03270878
Title: A Phase One, Single Dose, Randomized, Open-label, Two-period, Two-sequence, Crossover, Absolute Bioavailability Study Of Glasdegib (Pf-04449913) In Healthy Volunteers
Brief Title: Glasdegib Absolute Bioavailability Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B1371022
Record Dates: First submitted 2017-08-31; First posted 2017-09-01 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Healthy Volunteer Study
Keywords: Glasdegib; PF-04449913; Pharmacokinetics; Bioavailability
MeSH Terms: interventions — glasdegib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Glasdegib Oral tablet then IV (Experimental): Subjects will receive a single 100 mg oral tablet of glasdegib under fasted conditions in the first study period followed by washout. Then in the second period, a 50 mg IV solution will be infused over approximately 1.25 hours under fasted conditions.
  Interventions: Drug: Glasdegib Oral Tablet; Drug: Glasdegib IV infusion
- Glasdegib IV solution followed by Oral tablet (Experimental): Subjects will receive a 50 mg IV solution will be infused over approximately 1.25 hours in the fasted condition followed by washout in the first study period . Then in the second period, a single 100 mg oral tablet of glasdegib will be administered under fasted conditions
  Interventions: Drug: Glasdegib Oral Tablet; Drug: Glasdegib IV infusion

INTERVENTIONS:
Drug: Glasdegib Oral Tablet — Subjects will receive a single 100 mg oral tablet of glasdegib under fasted conditions, either in study period 1 or 2, depending on randomization.
Drug: Glasdegib IV infusion — Subjects will receive a 50 mg IV infusion of glasdegib over approximately 1.25 hours, in the fasted state, in either period 1 or 2 based on randomization.

SUMMARY:
This study is intended to estimate the absolute bioavailability of Glasdegib by comparison of the pharmacokinetic exposures following administration of an oral, single dose 100 mg tablet vs. an IV infusion of a 50 mg IV dose in the fasted state in a crossover fashion to healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:
* Healthy male and/or female subjects of non-child bearing potential who, at the time of screening, are between the ages of 18 and 55 years, inclusive. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG or clinical laboratory tests. Female subjects of nonchildbearing potential must meet at least 1 of the following criteria:

  1. Achieved postmenopausal status, defined as follows: cessation of regular menses for at least 24 consecutive months with no alternative pathological or physiological cause; with a serum follicle-stimulating hormone (FSH) level confirming the postmenopausal state;
  2. Have undergone a documented hysterectomy and/or bilateral oophorectomy;
  3. Have medically confirmed ovarian failure. All other female subjects (including females with tubal ligations and females that do NOT have a documented hysterectomy, bilateral oophorectomy and/or ovarian failure) are considered to be of childbearing potential.
* Body mass index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).
* Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study. -. Subjects who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* -A positive urine drug test.
* Screening supine 12-lead ECG demonstrating a corrected QT (QTc) interval >450 msec or a QRS interval >120 msec. If QTc exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated 2 more times and the average of the 3 QTc or QRS values should be used to determine the subject's eligibility.
* Subjects with family history of myocardial infarction, congenital long QT syndrome, torsades de pointes or clinically significant ventricular arrhythmias. Subjects should be within normal range of potassium, magnesium and corrected calcium calculation at screening.
* Pregnant female subjects; breastfeeding female subjects; female subjects of childbearing potential; male subjects with partners currently pregnant; male subjects who are unwilling or unable to use two highly effective methods of contraception as outlined in this protocol for the duration of the study and for at least 90 days after the last dose of investigational product and, refrain from sperm donation for the duration of the Study and for at least 90 days after the last dose of investigational product.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-09-07 (Actual); Primary Completion 2017-10-06 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
Dose Normalized Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - 8)] | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- New Haven Clinical Research Unit, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Information relating to our policy on data sharing and the process for requesting data can be found at the following link: http://www.pfizer.com/research/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Shaik N, Hee B, Liang Y, LaBadie RR. Absolute Oral Bioavailability of Glasdegib (PF-04449913), a Smoothened Inhibitor, in Randomized Healthy Volunteers. Clin Pharmacol Drug Dev. 2019 Oct;8(7):895-902. doi: 10.1002/cpdd.692. Epub 2019 Apr 12. PMID 30977980
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1371022&StudyName=A+Phase+One%2C+Single+Dose%2C+Randomized%2C+Open-label%2C+Two-period%2C+Two-sequence%2C+Crossover%2C+Absolute+Bioavailability+Study+Of+Glasdegib+%28pf-04449913%29+In+Healthy+Volunteers